CLINICAL TRIAL: NCT05196685
Title: Is Carotid-Vertebral Doppler Ultrasonography Necessary for Patients With Vertigo?
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Prof. Dr., Pamukkale University
Other Study IDs: 10
Record Dates: First submitted 2022-01-03; First posted 2022-01-19 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Vertigo; Carotid Artery Diseases
Keywords: Vertigo; Imbalance; Doppler Ultrasonography; Carotid Artery; Vertebral Artery
MeSH Terms: conditions — Vertigo; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Vertigo: Patients who have Carotid Doppler Ultrasonography and Vertigo screening test scores of 1 and above will be sent to ENT
  Interventions: Diagnostic Test: Carotid Doppler USG
- Group control: Patients who have Carotid Doppler Ultrasonography and Vertigo screening test score below 1
  Interventions: Diagnostic Test: Carotid Doppler USG

INTERVENTIONS:
Diagnostic Test: Carotid Doppler USG — All Doppler ultrasonography measurements will be made in a dimly lit room at room temperature, with the patient in the supine position, the head slightly hyperextended, the patient looking to the left when measuring the right side, and the patient looking to the right when measuring the left side. In all patients, common carotid artery (CCA), internal carotid artery (ICA) and vertebral artery (VA) gray scale and color Doppler ultrasonography wşll be performed using the GE 9L Linear Probe. Color Doppler examination will be performed with a frequency of 4.0/8.0 MHz.

SUMMARY:
This study will be carried out prospectively on patients who applied to the cardiovascular surgery polyclinic and the carotid-vertebral artery doppler ultrasound due to the vascular problem. All patients will fill "Balance Disorder Scan Survey" and "Vertigo-Dizziness Imbalance Questionnaire-SS". Patients who score 1 and more are directed to the ear nose throat polyclinic and detailed differential diagnosis. Those who score 0 will be in control group.

DETAILED DESCRIPTION:
Right and left carotid artery flow velocities, intima-media thicknesses (IMT), presence of plaque, vertebral artery flow velocities, and vertebral artery resistance indexes (RI) will be recorded in all patients. Risk factor analysis, Vertigo Symptom Scale (VSS) and Dizziness Handicap Inventory (DHI-S) questionnaires will be applied to the patients in the ENT outpatient clinic. The differential diagnosis of vertigo will be made by performing detailed balance examinations and advanced balance tests.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have a vascular problem and doppler USG.

Exclusion Criteria:

Patients with impaired cooperation, history of malignancy, presence of central nervous system pathology, presence of neurological disease affecting balance in the history, patients whose use of glasses may cause problems (epilepsy, vision loss, etc.) were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be conducted prospectively on patients who apply to the Cardiovascular Surgery outpatient clinic and undergo Carotid-vertebral artery Doppler ultrasound due to vascular problems.
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Carotid Stenosis | 1 year
  ECST for Carotid Stenosis measurement will be used. In the ECST the estimated normal lumen diameter at the site of the lesion, based on a visual impression of where the normal arterial wall is before development of the stenosis, is used.
Resistive Index | 1 year
  Measurements are taken from vertebral artery and formulated as below.
  Resistive Index = peak systolic velocity - end diastolic velocity] / peak systolic velocity
Intima Media Thickness | 1 year
  The intima-media thickness will be measured 1 cm proximal to the start of the carotid bulb dilatation on the CCA in the far wall. Using the cine-loop function, an optimal longitudinal freeze-frame image in the end-diastolic state is measured manually.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided